CLINICAL TRIAL: NCT03171103
Title: Systemic Lupus and Pregnancy Outcome in Benisuef Localities
Brief Title: Systemic Lupus and Adverse Pregnancy Outcome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Momen Zakaria Mohammed mohammed, assisstant lecturer, Beni-Suef University
Other Study IDs: 2505
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Systemic Lupus Erythematosus; Pregnancy Complications
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
prospective analytical study of all pregnant ladies with systemic lupus in Beni-suef localities

ELIGIBILITY:
Inclusion Criteria:

* all pregnant ladies with settled diagnosis of systemic lupus

  * all pregnant ladies who first diagnosed as systemic lupus during current pregnancy

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: All pregnant ladies in Beni-suef localities diagnosed as systemic lupus
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
maternal outcome | 3 years
  Number of patients who have abortion,preterm labor,preeclampsia,eclampsia,accidental hemorrhage,oligohydramnios

SECONDARY OUTCOMES:
fetal outcome | 3 years
  Number of patients who have abortion,prematurity,Intrauterine growth restriction,intrauterine fetal death,still birth,low birth weight,neonatal death

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided